CLINICAL TRIAL: NCT05517018
Title: COMPARISON OF SINGLE, DOUBLE LAYER AND PURSE STRING TECHNIQUE (TURAN TECHNIQUE) STUR TYPES IN TERMS OF THE FORMATION OF UTERINE NICH FOR CLOSING THE UTERUS DURING CESERIAN SECTION
Brief Title: UTERUS CLOSURE TECHNIQUES and Uterine Niche Formation
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Yıldız, MEDİCAL DOCTOR, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasaTREHmmh
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Uterus; Scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- single layer uterotomy: 53 women with a single-layer uterotomy while closing the uterus during Ceserian
- double layer uterotomy: 53 women with a double layer uterotomy while closing the uterus during Ceserian
- purse string uterotomy: 53 women with a purse string uterotomy tecnique had used while closing the uterus during Ceserian

SUMMARY:
We aimed to compare 3 different uterotomy suture techniques with each other and evaluate them in terms of niche formation.1- one layer 2- double layer 3- purse string (TURAN technique)

DETAILED DESCRIPTION:
It is thought that the formation of the uterine niche may be mostly due to the surgical technique.We aimed to compare 3 different uterotomy suture techniques with each other and evaluate them in terms of niche formation.1- one layer 2- double layer 3- purse string (TURAN technique).

ELIGIBILITY:
Inclusion Criteria:

* have a cesarean section necessity
* be over 18 years old
* being younger than 40

Exclusion Criteria:

* emergency cesarean section
* Being under 37 weeks pregnant
* multiple pregnancies
* having had uterine surgery
* uterine malformations

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Patients who need to have a cesarean section will be included in the study.participants will be randomly divided into 3 groups according to the cesarean section technique.During the cesarean section, the uterus will be closed using different techniques for each of the 3 groups.6 weeks after the operation, they will be called for control and evaluated in terms of niche formation. and rezidue myometrial tissue
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
the formation of a uterine niche | 6 weeks
  The formation of a niche will be considered a failure, while the absence of a niche will be considered a technical success.

CONTACTS AND LOCATIONS:
Overall Officials: elif yıldız, Principal Investigator — Gaziosmanpasa Research and Education Hospital
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No